CLINICAL TRIAL: NCT06646601
Title: A Preventive, Multidisciplinary Primary Care Intervention Organized Around a Therapeutic Garden: Acceptability to Patients Suffering from Cardio-neurovascular Pathology and to Those Involved in the Action.
Acronym: ArTERRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: RCAPHM23_0482
Record Dates: First submitted 2024-10-14; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Vascular Disease; Cardiovascular; Atrial Fibrillation (AF); Heart Failure NYHA Class II; Cardiomyopathies; Stroke, Ischemic; Hypertension Resistant to Conventional Therapy
MeSH Terms: conditions — Vascular Diseases; Atrial Fibrillation; Cardiomyopathies; Ischemic Stroke; Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multidisciplinary preventive action and questionnaries (Experimental): A 6-month multidisciplinary preventive intervention for each patient: gardening, adapted physical activity, nutritional workshops and questionnaries
  Interventions: Other: Intervention of prevention
- No intervention but questionnaries (No Intervention): Refuse the intervention and answers questionnaries about why

INTERVENTIONS:
Other: Intervention of prevention — A 6-month multidisciplinary preventive intervention for each patient: gardening, adapted physical activity, nutritional workshops.
  Arms: Multidisciplinary preventive action and questionnaries

SUMMARY:
A preventive, multidisciplinary primary care intervention organized around a therapeutic garden: Acceptability to patients suffering from cardio-neurovascular pathology and to those involved in the action.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old;
* living in the vicinity (+-20 km) of Gap, Laragne-Montéglin, Veynes and Clermont-Ferrand;
* having been invited to take part in the intervention by the caregivers of the medical structures
* suffering from an ALD based on CNAM medical criteria (stroke, AOMI, rhythm disorders, valvular heart disease, congenital heart disease, stage I and II heart failure), severe hypertension, chronic coronary disease)

Exclusion Criteria:

* heart failure based on CNAM medical criteria (ALD n°5) stage III and IV according to NYHA classification ;
* with a contraindication to physical activity ;
* living in an institution;
* unable to walk more than 100 m independently;
* Alzheimer's disease or other dementias based on CNAM medical criteria ;
* with an unlabelled cognitive impairment limiting comprehension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Acceptance rate of intervention | From enrollment to the end of treatment at 6 months
  Assessing the acceptability of a multidisciplinary intervention combining gardening activities, APA and nutrition workshops, organized around a therapeutic garden, by patients suffering from cardio-neurovascular pathologies and the interveners of the action.
Identification of the obstacles and facilitators for intervention | From enrollment to the end of treatment at 6 months
  Identify the obstacles and factors facilitating patients' initial adhesion to and commitment to the scheme, and those influencing the implementation of the action by those involved, i.e. the facilitators and caregivers involved.

SECONDARY OUTCOMES:
Assessing the impact of the intervention | From enrollment to the end of treatment at 6 months
  Assess the impact of the intervention on quality of life, adoption of new lifestyle habits (PA and Mediterranean diet), depressive symptoms and physical performance, taking into account any adverse effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Gap +/- 20 km, Gap, France

IPD SHARING:
Plan to Share IPD: Undecided